CLINICAL TRIAL: NCT07333963
Title: Application of Kinesiotaping as an Adjunctive Physiotherapeutic Method in the Surgical Management of Impacted Mandibular Third Molars
Brief Title: Adjunctive Kinesiotaping in Surgical Treatment of Impacted Mandibular Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BNW/NWN/0052/KB1/57/I/23
Record Dates: First submitted 2025-12-09; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Impacted Third Molar Tooth
Keywords: kinesiotaping, impacted teeth
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research group (Experimental): Group undergoing Kinesiotaping after the surgical procedure
  Interventions: Other: Kinesiotaping; Procedure: extraction of impacted third lower molar
- Control Group (Other): no kinesiotaping
  Interventions: Procedure: extraction of impacted third lower molar

INTERVENTIONS:
Other: Kinesiotaping — basic lymphatic KT application
  Arms: Research group
Procedure: extraction of impacted third lower molar — basic surgical extraction

SUMMARY:
PATIENT INFORMATION SHEET Participants are invited to take part in a clinical study involving surgical removal of an impacted lower wisdom tooth. Participation in this study is entirely voluntary.

The purpose of this study is to observe the healing process after wisdom tooth removal and to assess whether the use of elastic therapeutic tape placed on the skin (kinesiotaping) may support recovery.

SURGICAL PROCEDURE The procedure will be performed under local anesthesia and will include: - Administration of local anesthesia

* Incision of the gum
* Exposure of the impacted tooth and surrounding bone
* Removal of the tooth
* Cleaning of the surgical site - Placement of sutures After the surgery, standard post■operative instructions will be provided. STUDY PROCEDURE

After the surgical procedure, patients will be randomly assigned to one of two groups:

1. Standard post■operative care
2. Post■operative care combined with application of elastic therapeutic tape on the skin of the face and neck area If the participants are assigned to the tape group, the tape will be applied immediately after surgery by qualified medical personnel and will remain in place for several days.

FOLLOW■UP VISITS Participant will be asked to attend follow■up visits on specific days after the procedure to allow the medical team to assess healing. PAIN MANAGEMENT Participant will be allowed to take pain medication if necessary, following medical advice.

VOLUNTARY PARTICIPATION Participation in this study is voluntary. Participant may withdraw from the study at any time without giving a reason and without affecting participants medical care.

CONFIDENTIALITY All medical information collected during the study will be handled confidentially and used solely for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases (generally healthy patient)

Indication for surgical extraction of impacted lower third molars for:

orthodontic reasons

surgical reasons

prophylactic reasons

Age between 16 and 64 years

Written informed consent to participate in the study

Exclusion Criteria:

* Presence of chronic systemic diseases, including:

diabetes mellitus

hypertension

autoimmune diseases

Pharmacological treatment in the period preceding the surgery

Pregnancy

Substance abuse or dependence

Head and neck malignancies

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-14 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
postoperative pain intensity | 2 days post-surgery and 7 days post-surgery
  Postoperative pain intensity will be assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores indicate greater pain intensity.
Maximum Mouth Opening (MMO) | FinishBefore surgery, 2 days after surgery, and 7 days after surgery
  Maximum mouth opening will be measured using a caliper as the interincisal distance between the upper and lower incisors at maximum mouth opening.
Facial Soft Tissue Swelling | Before surgery, 2 days after surgery, and 7 days after surgery
  Facial swelling will be assessed using linear tape measurements between six predefined facial reference points. The sum of distances will be used for analysis.
Postoperative Analgesic Consumption | Day of surgery, 2 days after surgery, and 7 days after surgery
  The total number of ketoprofen 100 mg tablets taken by each participant will be recorded as a measure of postoperative analgesic demand.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersyteckie centrum stomatologii, Bytom, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided